CLINICAL TRIAL: NCT06927440
Title: Development and Implementation of a National Multicenter Registry for Pediatric End-Stage Heart Failure in China
Brief Title: National Multicenter Registry for Pediatric End-Stage Heart Failure in China
Status: Enrolling by invitation | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Principal Investigator, Lijun Fu, Director of the Department of Cardiology, Shanghai Children's Medical Center, Shanghai Jiao Tong University School of Medicine
Other Study IDs: 2023YFC2706201
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure; Children
Keywords: end-stage heart failure; pediatric
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- National Multicenter Cohort for Pediatric End-Stage Heart Failure in China: A prospective multicenter cohort study on pediatric end-stage heart failure (ESHF) in China focusing on multicenter, multidimensional comprehensive analysis of demographic characteristics, risk factors, treatment efficacy, etiologies, prognoses, complications

SUMMARY:
To establish a multicenter pediatric end-stage heart failure (ESHF) specialized disease data platform and promote its adoption across major children's medical centers nationwide. Based on this platform, conduct a national multicenter cohort study on specialized treatments for pediatric ESHF (including pharmacotherapy, ventricular assist devices, heart transplantation, etc.). This initiative will provide a foundational platform for advancing national clinical research on pediatric end-stage heart failure.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet any of the following criteria despite receiving optimal guideline-directed medical therapy (GDMT):

Severe and persistent heart failure symptoms [New York Heart Association (NYHA) Class III (advanced) or IV];

Significant cardiac dysfunction, defined as:

Left ventricular ejection fraction ≤30%

Isolated right ventricular failure

Non-operable severe valvular or congenital abnormalities

Persistently elevated B-type natriuretic peptide (BNP) or N-terminal pro-BNP (NT-proBNP) levels

Severe diastolic dysfunction or left ventricular structural abnormalities (based on ESC definitions for heart failure with preserved ejection fraction [HFpEF] and heart failure with mildly reduced ejection fraction [HFmrEF]);

Requirement of:

High-dose intravenous diuretics (or combination diuretic therapy) for pulmonary/systemic congestion, OR

Inotropic/vasoactive agents for low cardiac output, OR

Management of malignant arrhythmias Resulting in >1 unplanned hospital visits or admissions within the past 12 months;

Severely impaired mobility due to cardiac causes with either:

Inability to ambulate, OR

6-minute walk distance <300 m, OR

Peak oxygen consumption (PvO₂) <12-14 mL/kg/min. -

Exclusion Criteria:

Concurrent life-limiting systemic disorders

Structural cardiac lesions with indication for surgical/interventional correction -

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with end-stage heart failure (ESHF) receiving care at multiple Chinese tertiary referral centers
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Composite of cardiovascular death, heart transplantation, LVAD implantation or WHF hospitalization | From enrollment to the follow up at 1 year, 3 years, 5 years
  WHF hospitalization: The patient was hospitalized for worsening heart failure; LVAD: left ventricular assistant device

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Children's Medical Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Skibelund AK; ESC Scientific Document Group. 2023 Focused Update of the 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2023 Oct 1;44(37):3627-3639. doi: 10.1093/eurheartj/ehad195. No abstract available. PMID 37622666
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW; ACC/AHA Joint Committee Members. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2022 May 3;145(18):e895-e1032. doi: 10.1161/CIR.0000000000001063. Epub 2022 Apr 1. PMID 35363499